CLINICAL TRIAL: NCT02494843
Title: Dynamic Effects of Online HDF on Cardiac Function and Myocardial Perfusion Utilising Cardiac MRI (CAMRID)
Acronym: CAMRID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 14025
Record Dates: First submitted 2015-07-07; First posted 2015-07-10 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Other Postprocedural Cardiac Functional Disturbances; Myocardial Perfusion
MeSH Terms: interventions — Hemodiafiltration; Renal Dialysis; Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online haemodiafiltration (Active Comparator)
  Interventions: Other: online Hemodiafiltration; Other: Hemodialysis
- Haemodialysis (Active Comparator)
  Interventions: Other: online Hemodiafiltration; Other: Hemodialysis

INTERVENTIONS:
Other: online Hemodiafiltration — Effects of high efficiency online hemodiafiltration on cardiac structure, function and myocardial perfusion were compared with standard haemodialysis.
  Other Names: Hemodiafiltration
Other: Hemodialysis — Effects of high efficiency online hemodiafiltration on cardiac structure, function and myocardial perfusion were compared with standard haemodialysis.
  Other Names: Haemodialysis

SUMMARY:
The purpose of this study is to characterise, in detail, the cardiac structure, function and perfusion of those on haemodialysis and haemodiafiltration, comparing the two modalities to ascertain if haemodiafiltration provides relative myocardial protection compared to conventional haemodialysis.

DETAILED DESCRIPTION:
Trial Configuration: Non-blinded crossover pilot study Setting: Secondary care Sample size estimate: This is a pilot study therefore power calculations are not appropriate. A group size of 12 participants has been selected for feasibility.

Number of participants: 12 patients to complete study Description of interventions

* 6 sessions of conventional haemodialysis each lasting 4 hours
* 6 sessions of online haemodiafiltration each lasting 4 hours
* 2 sessions of Cardiac MRI each lasting 6 hours in total to take place around 6th session of dialysis Randomisation and blinding: This is an open study. Statistical methods: All continuous variables will be tested for normality. The primary and continuous secondary endpoints will be compared between the two modalities using a paired t test or Wilcoxon signed rank test as appropriate. The association between categorical variables will be tested using the Chi squared or Fischer's Exact test. An alpha error at 0.05 will be judged as significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Able to give informed consent
* CKD5 on chronic haemodialysis
* Receiving dialysis via an arteriovenous fistula
* Must be able to follow simple instruction in English (on safety grounds for MRI scans)

Exclusion Criteria:

* Change in ideal dry weight in 4 weeks prior to recruitment
* Instability on dialysis in 4 weeks prior to recruitment leading to either:

  * Emergency medical attention
  * Infusion of additional fluid
  * Loss in consciousness
  * Arrhythmia
  * Chest pain
* Dialysed via a synthetic line or graft
* Qa < 500ml/min
* NYHA Stage IV heart failure
* Active infection or malignancy
* Contraindication to MRI scanning including claustrophobia
* Mental incapacity to consent
* Pregnancy or planning pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
The change in global cardiac perfusion (ml/min/100g) between conventional HD and HDF | 2 week

SECONDARY OUTCOMES:
The change in segmental cardiac perfusion during conventional HD and HDF | 2 week
The change in global and segmental cardiac function as measured by phase-contrast MRI | 2 week
Serum markers of cardiac damage, renal, liver function, clotting, full blood count | 2 weeks
  Bloods collected at the end of 2 week study period on the scan days on HD and HDF
Reported tolerability of cardiac MRI scanning whilst having dialysis | On 2 MRI study days
  On 2 MRI study days